CLINICAL TRIAL: NCT03205475
Title: JASPER Implementation Cascade: Newfoundland and Labrador
Brief Title: JASPER Implementation in NFLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Government of Newfoundland and Labrador (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GovernmentNL
Record Dates: First submitted 2017-06-27; First posted 2017-07-02 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Autism Spectrum Disorder
Keywords: Training; Intervention; Social Communication; Play
MeSH Terms: conditions — Autism Spectrum Disorder; Communication | interventions — Clinical Trials, Phase I as Topic

STUDY DESIGN:
Intervention Model Description: JASPER (Joint Attention, Symbolic Play, Engagement, and Regulation) is a play based targeted social communication intervention. Sessions will be delivered one on one by an interventionist in training with a child age 2.0-8.11 years who has autism.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- A. Above Fidelity Phase 1 and Above Fidelity Phase 2 (Active Comparator): Alternating coaching and streamed or video feedback each week through phase 1, moves to video feedback only for phase 2.
  Interventions: Behavioral: Alternate Coaching and Video Feedback Phase 1; Behavioral: Video Feedback Only Phase 2
- B. Below Fidelity Phase 1 and Above Fidelity Phase 2 (Active Comparator): Receive weekly coaching in phase 1, move to video feedback only in phase 2
  Interventions: Behavioral: Weekly Coaching in Phase 1; Behavioral: Video Feedback Only Phase 2
- C. Above Fidelity Phase 1, Below in Phase 2- Add Refresher (Active Comparator): Alternating coaching and streamed or video feedback each week through phase 1. In phase 2, the interventionist is still working toward 90% fidelity and is randomly assigned (50/50) to one of two different types of support from the Senior Trainer. The interventionist will receive a one week intensive in person refresher and then continue with weekly coaching and video feedback from the Senior Trainer (Enhanced Feedback plus intensive refresher course) for the final 12 weeks.
  Interventions: Behavioral: Alternate Coaching and Video Feedback Phase 1; Behavioral: Weekly Coaching plus Intensive Refresher Course Phase 2
- D. Above Fidelity Phase 1, Below in Phase 2- Add Peer (Active Comparator): Alternating coaching and streamed or video feedback each week through phase 1. In phase 2, the interventionist is still working toward 90% fidelity and is randomly assigned (50/50) to one of two different types of support from the Senior Trainer. The interventionist will receive weekly coaching and video feedback from the Senior Trainer plus a weekly session paired with a local interventionist at fidelity (Enhanced Feedback plus peer support).
  Interventions: Behavioral: Alternate Coaching and Video Feedback Phase 1; Behavioral: Weekly Coaching plus Peer Coaching Phase 2
- E. Below Fidelity Phase 1, Below in Phase 2- Add Refresher (Active Comparator): Receive weekly coaching in phase 1. In phase 2, the interventionist is still working toward 90% fidelity and is randomly assigned (50/50) to one of two different types of support from the Senior Trainer. The interventionist will receive a one week intensive in person refresher and then continue with weekly coaching and video feedback from the Senior Trainer (Enhanced Feedback plus intensive refresher course) for the final 12 weeks.
  Interventions: Behavioral: Weekly Coaching in Phase 1; Behavioral: Weekly Coaching plus Intensive Refresher Course Phase 2
- F. Below Fidelity Phase 1, Below in Phase 2- Add Peer (Active Comparator): Receive weekly coaching in phase 1. In phase 2, the interventionist is still working toward 90% fidelity and is randomly assigned (50/50) to one of two different types of support from the Senior Trainer. The interventionist will receive weekly coaching and video feedback from the Senior Trainer plus a weekly session paired with a local interventionist at fidelity (Enhanced Feedback plus peer support).
  Interventions: Behavioral: Weekly Coaching in Phase 1; Behavioral: Weekly Coaching plus Peer Coaching Phase 2

INTERVENTIONS:
Behavioral: Alternate Coaching and Video Feedback Phase 1 — Alternates each week between live/tele-health coaching (coaching) or Video review and call (feedback)
  Arms: A. Above Fidelity Phase 1 and Above Fidelity Phase 2; C. Above Fidelity Phase 1, Below in Phase 2- Add Refresher; D. Above Fidelity Phase 1, Below in Phase 2- Add Peer
Behavioral: Weekly Coaching in Phase 1 — Weekly coaching (live or telehealth)
  Arms: B. Below Fidelity Phase 1 and Above Fidelity Phase 2; E. Below Fidelity Phase 1, Below in Phase 2- Add Refresher; F. Below Fidelity Phase 1, Below in Phase 2- Add Peer
Behavioral: Weekly Coaching plus Intensive Refresher Course Phase 2 — Continue weekly coaching with senior trainer and add one week intensive refresher course
  Arms: C. Above Fidelity Phase 1, Below in Phase 2- Add Refresher; E. Below Fidelity Phase 1, Below in Phase 2- Add Refresher
Behavioral: Weekly Coaching plus Peer Coaching Phase 2 — Continue weekly coaching with senior trainer and add weekly peer coaching from another interventionist in the region who is at high fidelity
  Arms: D. Above Fidelity Phase 1, Below in Phase 2- Add Peer; F. Below Fidelity Phase 1, Below in Phase 2- Add Peer
Behavioral: Video Feedback Only Phase 2 — Receive video feedback and calls only
  Arms: A. Above Fidelity Phase 1 and Above Fidelity Phase 2; B. Below Fidelity Phase 1 and Above Fidelity Phase 2

SUMMARY:
This study will focus on examining the supports required to enable community Senior JASPER Trainers to support the training and development of junior interventionists throughout the province of Newfoundland and Labrador, Canada. The study will examine the training and supports delivered by Senior Trainers to help junior interventionists provide a targeted social communication intervention (JASPER: Joint Attention, Symbolic Play, Engagement, and Regulation) with children with autism spectrum disorder (ASD). Children's engagement, play, and social communication outcomes will be examined as well as the influence of junior interventionists' intervention implementation on children's outcomes. Further, the study will examine the supports required to help junior interventionists who demonstrate slower gains in implementation fidelity after the first three months of standard support. Interventionists who are slow to gain implementation fidelity will be randomized to either (a) enhanced feedback plus peer support or (b) enhanced feedback plus intensive refresher course.

DETAILED DESCRIPTION:
The proposed study is an adaptive intervention trial that will focus on tailoring supports for new JASPER interventionists. Coaching and training supports will be provided by Local Senior JASPER Trainers will support the development of new interventionists. Based on the interventionist's individual response to the coaching/training supports, a change in support may be provided at a priori time points including end of month 1 (training case) if at least 70% fidelity is not reached, and at end of month 4 (midpoint of first child cohort), at least 90% fidelity is not reached.

ELIGIBILITY:
Inclusion Criteria:

* Children: Must be 2.0-8.11 years of age; must meet the scoring benchmark for "autism" or "autism spectrum disorder" on the ADOS-2; has not previously received JASPER intervention in the province
* Interventionists: Work as an interventionist for the Government of Newfoundland and Labrador; minimum educational requirement is a Bachelor's Degree or Master's Degree in Psychology or a related field
* Senior JASPER Trainers: - Have been trained previously in JASPER; Work as a Senior Trainer for the Government of Newfoundland and Labrador; Minimum educational requirement is a Master's degree in a related field (e.g., Speech and Language Pathology, Occupational Therapy, Developmental Psychology).

Exclusion Criteria:

* Children: Child is below 2.0 years of age or above 8.11 years of age; Child does not meet the benchmark for autism or autism spectrum disorder on the ADOS-2; Child has received JASPER intervention prior to this study
* Interventionists: Not employees of the Government of Newfoundland and Labrador; does not hold a Bachelor's degree in a related field
* Senior Trainers: No prior JASPER training; Not employees of the Government of Newfoundland and Labrador; does not hold a Master's Degree in a related field

Ages: 24 Months to 97 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Change in JASPER Strategy Implementation Fidelity | Entry, 1 month, 4 months, and 7 month exit
  Quantitative ratings of the interventionists' quality and accurate use of JASPER intervention strategies.

SECONDARY OUTCOMES:
Change in Children's Joint Engagement | Entry for cohort two (month 2), half way (month 4), and exit (month 7)
  Time the child spends jointly engaged in interactions with the interventionist
Change in Children's Play Skills and Social Communication Skills | Entry for cohort two (month 2), half way (month 4), and exit (month 7)
  Rated during the child's interactions with the interventionist and during independent assessment, this includes the child's spontaneous play types by play level and child's spontaneous spoken and nonverbal communication skills to request and to share

CONTACTS AND LOCATIONS:
Overall Officials: Connie Kasari, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Department of Health and Community Services, Government of Newfoundland and Labrador, St. John's, Newfoundland and Labrador, Canada

IPD SHARING:
Plan to Share IPD: No